CLINICAL TRIAL: NCT05220306
Title: AIDI - Research & Development of a Multisensor-Based Machine Learning Technology for Real-Time Automated Detection of COVID-19 Decompensation
Acronym: AIDI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No eligible patients could be found and funding was lost
Sponsor: AIDAR Health, Inc. (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: ADR04-AIDI-C-21
Record Dates: First submitted 2022-02-01; First posted 2022-02-02 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-02

CONDITIONS: Sars-CoV-2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Phase I/Derivation Cohort (100 patients):
  This phase will use the MouthLab to capture vital signs. This data will help create Aidar's algorithm-based decompensation index (AIDI) that utilizes changes in vital signs to identify individuals who test positive for SARS-CoV-2 or with COVID-19 infection and are at risk of developing clinical decompensation.
  Phase II/Validation Cohort (400 patients):
  This phase will use the MouthLab to capture vital signs and use Aidar's algorithm-based decompensation index (AIDI) to identify individuals at risk of clinical decompensation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Device Arm (Experimental): Participants will use the MouthLab device for monitoring their vital signs
  Interventions: Device: Monitoring of vital signs

INTERVENTIONS:
Device: Monitoring of vital signs — The MouthLab is a hand-held device. The user holds the unit in their left hand with the Mouthpiece between the teeth and lips and breathes normally into the device for 30 seconds.

SUMMARY:
The AIDI study has to phases. It's purpose is to capture vital signs using a non-invasive, hand-held, home monitoring device (MouthLab Device) from individuals with COVID-19 or who test positive for SARS-CoV-2 (Phase I) and use an algorithm-based approach to identify individuals at risk of clinical decompensation (Phase II). Up to 500 unvaccinated and partially vaccinated subjects will be included (up to 100 in Phase I and up to 400 in Phase II).

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age or older
* Unvaccinated individuals, or individuals who have received only 1 dose of an mRNA vaccine
* Individuals who have received a positive SARS-CoV-2 result within 24-48 hours (lab-based PCR or antigen test)
* Willing and able to provide informed consent
* Ability to read, write, and comprehend English
* Have no functional limitation that would impede the use of the MouthLab device
* Willing to provide access to health information via electronic health records (EHR)

Exclusion Criteria:

* Currently receiving hospice care
* Have a left ventricular assist device
* Left-sided hemiplegia or any other motor deficits that may restrict the use of the device.
* individuals with cognitive deficits that impede their ability to comprehend and give informed consent.
* Individuals who are enrolled in any other investigational research studies of SARS-CoV2 or COVID-19
* Individuals who are treated with monoclonal antibody therapy prior to diagnosis
* Individuals who are admitted to a hospital or acute care facility at the time of diagnosis
* Individuals with pacemakers or implanted cardio-defibrillators (ICDs)
* History of hemoptysis, pneumothorax, thoracic or abdominal aneurysm, pulmonary embolism, or stroke
* History of unstable cardiovascular status, including recent myocardial infarction (MI within 30 days), unstable angina, or uncontrolled hypertension Color blindness
* Chest, abdominal or eye surgery within the preceding 14 days
* Any condition that in the judgment of the investigators would interfere with the subject's ability to provide informed consent, comply with study instructions, place the subject at increased risk, or which might confound interpretation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Collect trends in physiological vital signs and symptom burden to identify individuals who are at risk of clinical decompensation | Daily for 60 days
  Accurately collect trends in physiological vital signs and symptom burden of individuals with COVID-19 infection or who test positive for SARS-CoV-2 captured with the MouthLab to identify individuals who are at risk of clinical decompensation. (Phase 1)
AIDI evaluation | Daily for 60 days
  Evaluate trends in physiological vital signs and symptom burden of individuals with COVID-19 infection or who test positive for SARS-CoV-2 which are captured with the MouthLab device to evaluate the ability of the Aidar COVID-19 Decompensation Index (AIDI) to accurately identify individuals at risk of clinical decompensation. (Phase 2)

SECONDARY OUTCOMES:
Usability of MouthLab device | At 60 days
  Usability of the MouthLab device will be assessed via a questionnaire at study exit
Evaluate any short-term changes in vital signs among patients with underlying comorbid conditions | Day 0 to Day 60
  Evaluate any short-term changes in vital signs among patients with underlying comorbid conditions

CONTACTS AND LOCATIONS:
Overall Officials: Sujith Shetty, MD, Principal Investigator — Avania
Locations (1):
- Maxis Llc, San Jose, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mathew J, Pagliaro JA, Elumalai S, Wash LK, Ly K, Leibowitz AJ, Vimalananda VG. Developing a Multisensor-Based Machine Learning Technology (Aidar Decompensation Index) for Real-Time Automated Detection of Post-COVID-19 Condition: Protocol for an Observational Study. JMIR Res Protoc. 2025 Mar 27;14:e54993. doi: 10.2196/54993. PMID 40146983